CLINICAL TRIAL: NCT02015741
Title: Comparability of Bispectral Index and NeuroSENSE in Aged Patients
Status: Withdrawn | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/36; 2012-A01192-41 (Other: ANSM)
Record Dates: First submitted 2013-12-05; First posted 2013-12-19 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Sleep
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aged patients: EEG monitoring with Bispectral Index and NeuroSENSE
  Interventions: Device: EEG monitoring with Bispectral Index and NeuroSENSE; Behavioral: Clinical observation

INTERVENTIONS:
Device: EEG monitoring with Bispectral Index and NeuroSENSE
Behavioral: Clinical observation — Patients will be observed during awake periods and during natural sleep.

SUMMARY:
The assessment of anesthesia depth was based, until recently, on the evolution of hemodynamic parameters. Nowadays it can be evaluated by several monitoring methods, derived from electroencephalogram analysis, namely the Bispectral Index (Aspect Medical Systems, Newton, USA). A new modality is currently under development: the NeuroSENSE (Cleveland Medical Devices Inc., Cleveland, OH 44103, USA).

Use of such devices is discussed in aged patients. The purpose of this study is to compare Bispectral Index and NeuroSENSE during awake periods and during natural sleep.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 74 years

Exclusion Criteria:

* pace-maker

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Aged patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a high concordance between pairs of Bispectral Index and NeuroSENSE indices | 1 year
  Statistical analysis of concordance between pairs of Bispectral Index and NeuroSENSE indices (high concordance when > 0.60%)

SECONDARY OUTCOMES:
Percentage of patients with a high concordance between pairs of Bispectral Index and NeuroSENSE indices during periods of natural sleep | 1 year
  Statistical analysis of concordance between pairs of Bispectral Index and NeuroSENSE indices measured during periods of natural sleep (high concordance when > 0.60%)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bresson, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Hopital Stell, Rueil, Hauts de Seine
  - Hopital Foch, Suresnes, Hauts de Seine